CLINICAL TRIAL: NCT00678132
Title: A Phase I Combination Study of AZD2281 and Cisplatin Plus Gemcitabine in Adults With Solid Tumors
Brief Title: AZD2281 and Cisplatin Plus Gemcitabine to Treat Solid Tumor Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080128; 08-C-0128; NCT01445457 (obsolete NCT alias)
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2012-09-07

CONDITIONS: Neoplasms
Keywords: PARP Inhibitor; Combination Study; Chemotherapy; Advanced Cancer; Neoplasms; Cancer; Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — olaparib; Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: AZD 2281
Drug: Cisplatin
Drug: Gemcitabine

SUMMARY:
Background:

* AZD2281 is an experimental drug in a class of agents called PARP inhibitors. PARP is a protein that is involved in repairing DNA damage; PARP inhibitors interfere with that process.
* Cisplatin and gemcitabine are approved by the United States Food and Drug Administration to treat certain cancers.

Objectives:

* To determine the optimum doses of AZD2281, cisplatin and gemcitabine in combination that can safely be given to patients with solid tumor cancers.
* To evaluate the response of the tumor to the drug combination and determine the side effects of the treatment.

Eligibility:

-Patients 18 years or older with an advanced solid tumor cancer for whom standard treatments are not effective.

Design:

* In this dose escalation study, the first small group of patients receives the smallest study doses of the study drugs. Subsequent groups receive incrementally higher doses as long as the preceding group does not experience unacceptable side effects. When the highest safe dose is determined, additional patients entering the study receive that dose.
* Patients receive treatment in 21-day cycles as follows:
* Days 1-4: AZD2281 by mouth twice a day
* Day 3: gemcitabine thorough a vein over 1 hour; then cisplatin through a vein over 1 hour.
* Day 10: gemcitabine through a vein over 1 hour.
* Evaluations during treatment include the following:
* Physical examination, vital signs check and blood tests every 3 weeks.
* CT scans every 6 weeks to evaluate the tumor.
* Treatment may continue until it is no longer beneficial.

DETAILED DESCRIPTION:
Background:

* Poly (ADP-ribose) polymerase-enzyme (PARP-1) recognizes and rapidly binds to DNA single- and double-strand breaks and has been shown to participate in other DNA-related functions, including gene amplification, cell division, differentiation, apoptosis, and DNA base-excision repair.
* Increased PARP activity is one of the mechanisms by which tumor cells avoid apoptosis caused by DNA damaging agents, and drug resistance has been linked to higher expressions of PARP in cancer cells. This differential expression of PARP supports the observed selectivity of PARP inhibitors to affect proliferating tumor cells. AZD2281 is an orally administered potent inhibitor of PARP-1 and PARP-2, and its combination with cisplatin and gemcitabine may overcome some of the resistance associated with these agents.

Primary Objectives:

* Establish the safety, tolerability, and maximum tolerated dose (MTD) of AZD2281 in combination with cisplatin and gemcitabine in patients with solid tumors.
* Evaluate the effect of cisplatin-gemcitabine, with or without AZD2281, on PAR and gamma- H2AX levels in tumor biopsies and peripheral blood mononuclear cells (PBMCs) pre- and post-treatment.

Secondary Objectives:

- Evaluate the pharmacokinetics (PK) of AZD2281 with and without cisplatin and gemcitabine.

Eligibility:

* Patients (greater than or equal to 18 years) must have histologically confirmed solid tumor malignancy that is metastatic or unresectable for which standard curative measures do not exist, or are associated with minimal patient survival benefit.
* Patients who have previously received cisplatin or gemcitabine, or both, are eligible.

Design:

* Cycle 1 and subsequent cycles: AZD2281 will be administered orally every 12 hours (Q 12 hours) on day 1, while gemcitabine will be administered intravenously (IV) over 1 hour (600 mg/m(2)/hour) on day 1 and 8 of each cycle and cisplatin over 1 hour on day 1 after gemcitabine.
* Dose escalation will proceed in cohorts of 3 6 patients to a minimum of 27 and a maximum of 42 patients.
* Patients will have a maximum of six cycles of treatment.
* Tumor biopsies will be collected in cycle 1 only, while blood for PBMC samples will be collected in cycle 1 and before drug administration, 24 and 48 hours post administration, in cycle 2, day 1. If Dose Level 3 is achieved additional time points will be collected in cycle 1, day 8 - before drug administration, 6, 24 and 48 hours

post.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histologically confirmed (by the NIH pathology department) solid tumor malignancy that is metastatic or unresectable for which standard curative measures do not exist, or are associated with minimal patient survival benefit.

* To minimize the risk of bone marrow toxicity in this population, patients must have had no more than two prior severely myelosuppressive cytotoxic chemotherapy regimens.
* Any prior therapy must have been completed greater than 2 weeks prior to enrollment on the protocol in patients participating in a phase 0 (eIND]) study, or greater than or equal to 4 weeks in patients participating in a regulatory IND study, and the participants must have recovered to eligibility levels (CTCAE Grade less than or equal to 1) from prior toxicity. Prior radiation or surgery should have been completed greater than or equal to 4 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels (prior irradiated tumors will be considered for biopsy if signs of disease progression are present).
* Age greater than or equal to18 years. Because no dosing or AE data are currently available on the use of AZD2281 in patients less than 18 years of age, children are excluded from this study, but may be eligible for future pediatric Phase I combination trials.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60 percent).
* Life expectancy greater than or equal to 3 months.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/microL
  * Platelets greater than or equal to 100,000/microL
  * Total bilirubin less than or equal to 1.5 times institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 times institutional upper limit of normal
  * Creatinine less than or equal to 1.5 times institutional upper limit of normal

OR

* Creatinine clearance greater than or equal to 60 mL/minute for patients with creatinine levels greater than 1.5 times institutional upper limit of normal.

  * The effects of AZD2281 on the developing human fetus are unknown. For this reason, and because cisplatin and gemcitabine used in this trial are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after completion of study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
  * Ability to understand and the willingness to sign a written informed consent document.
  * Patients who have previously received cisplatin or gemcitabine, or both, are eligible to enter the trial.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study, or those who have not recovered from AEs due to agents administered more than 4 weeks earlier. Patients must be greater than or equal to 2 weeks since any investigational agent was administered as part of an exploratory IND study and should have recovered to eligibility levels from any toxicity.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, prolonged QTc interval (greater than 500 msec), or psychiatric illness/social situations that would limit compliance with study requirements.
* In the Food and Drug Administration (FDA) Use-in-Pregnancy Ratings for Drugs, cisplatin and gemcitabine are classified as category D drugs, indicating that investigational or postmarketing data show risk to the fetus. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after completion of study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is a risk for AEs in nursing infants secondary to treatment of the mother with these drugs, breastfeeding should be discontinued while the patient is on this trial and for 30 days after completion of treatment on this trial.
* Patients with known brain metastases are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status remains stable for greater than or equal to 1 month after treatment of the brain metastases without steroids (except for maintenance replacement doses of steroids) or anti-seizure medications.
* Patients with clinically significant illnesses which could compromise participation in the study, including, but not limited to, active or uncontrolled infection, immune deficiencies or confirmed diagnosis of HIV infection, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are excluded from this trial.
* Patients with lymphomas and primary CNS malignancies are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04-24; Primary Completion 2010-11-23 (Actual); Study Completion 2010-11-23 (Actual)

PRIMARY OUTCOMES:
Establish the safety and tolerability of AZD2281 in combination with cisplatin and gemcitabine in patients with solid tumors. Establish the maximum tolerated dose (MTD) for the combination of AZD2281 with cisplation and gemcitabine.

SECONDARY OUTCOMES:
Evaluate the effect of chemotherapy (cisplatin-gemcitabine) with or without AZD2281 on PAR levels and g-H2AX levels in tumor biopsies and peripheral blood mononuclear cells (PBMCs) pre- and post treatment. Evaluate the pharmacokinetic (PK) of A.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ame JC, Spenlehauer C, de Murcia G. The PARP superfamily. Bioessays. 2004 Aug;26(8):882-93. doi: 10.1002/bies.20085. PMID 15273990
- [Background] D'Amours D, Desnoyers S, D'Silva I, Poirier GG. Poly(ADP-ribosyl)ation reactions in the regulation of nuclear functions. Biochem J. 1999 Sep 1;342 ( Pt 2)(Pt 2):249-68. PMID 10455009
- [Background] d'Adda di Fagagna F, Hande MP, Tong WM, Lansdorp PM, Wang ZQ, Jackson SP. Functions of poly(ADP-ribose) polymerase in controlling telomere length and chromosomal stability. Nat Genet. 1999 Sep;23(1):76-80. doi: 10.1038/12680. PMID 10471503
- [Derived] Shamseddine AI, Farhat FS. Platinum-based compounds for the treatment of metastatic breast cancer. Chemotherapy. 2011;57(6):468-87. doi: 10.1159/000334093. Epub 2012 Jan 10. PMID 22248721